CLINICAL TRIAL: NCT01115595
Title: Efficacy of Mite Allergen Vaccine Among Thai Patients With Allergic Rhinitis
Brief Title: Efficacy of Allergen Immunotherapy for Allergic Rhinitis in Thais
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pongsakorn Tantilipikorn (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor-Investigator, Pongsakorn Tantilipikorn, Associate Professor Dr., Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 336/2552
Record Dates: First submitted 2010-05-01; First posted 2010-05-04 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Allergic rhinitis; Allergen injection immunotherapy; Efficacy
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): injection by Mite extract with standard allergic medication (oral antihistamine and/or topical nasal steroid)
  Interventions: Biological: Intervention
- Control Group (Other): Injection by buffer solution WITH standard allergic medication (oral antihistamine and/or topical nasal steroid
  Interventions: Other: Control

INTERVENTIONS:
Biological: Intervention — Dermatophagoides pteronyssinus from ALK company
  Other Names: Mite allergen extract (D.p) from ALK company. 10,000 AU/ml
  Arms: Intervention
Other: Control — Injection by buffer solution WITH standard allergic medication (oral antihistamine and/or topical nasal steroid)
  Arms: Control Group

SUMMARY:
The purpose of this study is to study the efficacy of allergen injection immunotherapy for allergic rhinitis by

* symptoms score
* medication score
* quality of life
* immunologic test from blood

DETAILED DESCRIPTION:
Compare the efficacy of allergen injection immunotherapy between the treatment group and the placebo group after injection for

* 2 months
* 6 months
* 12 months

ELIGIBILITY:
Inclusion Criteria:

* patients with the symptoms of allergic rhinitis who sensitized to mite (Dermatophagoides pteronyssinus)
* positive skin prick test to D.p. at 4+ degree

Exclusion Criteria:

* steroid dependent asthma
* force expiratory volume (FEV1) less than 70% of predicted value
* previous injection immunotherapy within 2 years
* pregnancy
* medical conditions such as ischemic heart disease, autoimmune disease, cancer, previous history of anaphylaxis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-03; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Total nasal symptoms score | average within 1 week
  3 point scale (0,1,2,3) and combination of
  * nasal block
  * rhinorrhea
  * itching
  * sneezing

SECONDARY OUTCOMES:
Combined total symptoms score and medication score | average within 1 week
  Total symptom score (nasal block, rhinorrhea, itching, sneezing, and eye symptoms with chest symptoms = Maximal score --> 18 devided by 6 = 3) PLUS medication score ( antihistamine = 1, topical nasal steroid = 2; --> Maximal score = 3).

CONTACTS AND LOCATIONS:
Overall Officials: Pongsakorn Tantilipikorn, M.D., Principal Investigator — Division of allergy and rhinology, Faculty of Medicine Siriraj, Mahidol University
Locations (1):
- Division of Allergy and Rhinology, Faculty of Medicine Siriraj, Mahidol University, Bangkok, Thailand